CLINICAL TRIAL: NCT02073838
Title: A Phase II, Multi-center, Open Label, Randomized Study of Ribavirin and Hedgehog Inhibitor With or Without Decitabine in Acute Myeloid Leukemia (AML)
Brief Title: Ribavirin and Hedgehog Inhibitor With or Without Decitabine in AML
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sarit Assouline (Other)
Responsible Party: Sponsor-Investigator, Sarit Assouline, Hematologist-oncologist, Jewish General Hospital
Organization: Jewish General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ribavirin=005
Record Dates: First submitted 2014-02-21; First posted 2014-02-27 (Estimated); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Ribavirin; HhAntag691; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ribavirin, vismodegib, decitabine (Experimental): Decitabine 20mg/m2 IV QD days -7 to -3 for cycle 1. Ribavirin 1400mg BID and vismodegib 150mg QD starting on day 1. On subsequent cycles, decitabine will be administered on days 1 to 5.
  Interventions: Drug: Ribavirin; Drug: Vismodegib; Drug: Decitabine
- Ribavirin, vismodegib (Experimental): Ribavirin 1400mg BID, vismodegib 150mg QD
  Interventions: Drug: Ribavirin; Drug: Decitabine

INTERVENTIONS:
Drug: Ribavirin
Drug: Vismodegib
  Arms: Ribavirin, vismodegib, decitabine
Drug: Decitabine

SUMMARY:
This is a research study of ribavirin which will be given in combination with vismodegib and/or decitabine. The purpose of this study is to see if patients respond to treatment when ribavirin is given with vismodegib alone or in combination with decitabine.

ELIGIBILITY:
INCLUSION CRITERIA

1. Patients with AML M4 or M5 FAB subtype or high eIF4E are eligible.
2. All patients must have failed primary therapy (defined as two induction chemotherapies), must have relapsed, or must not be suitable candidates for intensive induction chemotherapy.
3. Patients who have a dry aspirate or extramedullary disease only are eligible for this study if they have a pre-treatment marrow or tissue biopsy demonstrating AML M4 or M5 subtype or high eIF4E.
4. ECOG performance status 0, 1, 2.
5. Life expectancy>4 weeks.
6. Age is > 18 years.
7. Female patients of childbearing potential (FCBP) is defined as a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy, or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months). In addition, women under the age of 55 years must have a serum follicle stimulating hormone (FSH) level > 40IU/L to confirm menopause.

   FCBP must have a negative serum (beta-HCG) pregnancy test (minimum sensitivity 25 IU/L of equivalent units of HCG) within 7 days of starting treatment and must not be breastfeeding. Men and females of childbearing potential must agree to use two effective means of contraception, with one method being highly effective and the other method being either highly effective or less effective as listed below throughout the study and for at least 24 months after completion of protocol.

   An effective means of contraception includes the following:

   i. Male condoms with spermicide ii. Hormonal methods of contraception including combined oral contraception pills, vaginal ring, injectables, implants, and intrauterine devices (IUDs).

   iii. Nonhormonal IUDs iv. Tubal ligation v. Vasectomy vi. Complete Abstinence

   A less effective means of contraception includes the following:

   i. Diaphragm with spermicide ii. Vaginal sponge iii. Male condom without spermicide iv. Progestin only pills by females of childbearing potential or male subject's FCBP partners v. Female condom (a male and female condom must not be used together)

   Male subjects must not donate semen while on study and during 24 months after treatment discontinuation.
8. Adequate renal and hepatic function: serum creatinine < 1.5 x ULN; AST or ALT < 2.5 x ULN (or < 5 x ULN if liver involvement with leukemia); serum bilirubin < 1.5 x ULN
9. Provide written consent after the investigational nature, study design, risks and benefits of the study have been explained.
10. Accessible for treatment and follow up.

EXCLUSION CRITERIA

1. Patients with impaired ribavirin uptake. As tested in the central laboratory.
2. Uncontrolled central nervous system involvement by AML.
3. Active cardiovascular disease as defined by New York Heart Association (NYHA) class III-IV categorization.
4. Patients with hemoglobinopathies which may affect their ability to tolerate ribavirin.
5. Intercurrent illness or medical condition precluding safe administration of the planned protocol treatment or required follow-up.
6. Received any previous therapy for AML within 28 days prior to the study entry. Hydrea is permitted for the treatment of leukocytosis but must be stopped prior to starting study drugs.
7. Female patients who are pregnant or breastfeeding.
8. Concurrent treatment with other anti-cancer therapy except adjuvant antihormonal agents for breast cancer or for limited stage prostate cancer.
9. Known infection with HIV.
10. History of other active malignancy. Subjects who have been disease-free for 2 year or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible.
11. FAB AML M1, 2, 6, 7 will be excluded if they do not have high eIF4E expression. AML M3 is always excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2022-11 (Actual); Study Completion 2022-11 (Actual)

PRIMARY OUTCOMES:
Efficacy will be measured by overall response rate (ORR). | Measured up to 2 years after the last subject has enrolled in the study.

SECONDARY OUTCOMES:
Time to response | Measured up to 2 years after the last subject has enrolled in the study.
Duration of response | Measured up to 2 years after the last subject has enrolled in the study.
One year survival | Measured up to 2 years after the last subject has enrolled in the study.
Overall survival | Measured up to 3 years after the last subject has enrolled in the study.
Hematologic improvement defined by the number of individual, positively affected cell lines (erythroid, neutrophil and platelet cells) per patient. | Measured up to 2 years after the last subject has enrolled in the study.
Number of participants with Adverse Events as a Measure of Safety and Tolerability | Measured up to 2 years after the last subject has enrolled in the study.
Changes in eIF4E expression, localization, and signalling pathways (measured by immuno-histochemical analysis, PCR or western blot) and correlating with each patient's overall response. | Measured up to 2 years after the last subject has enrolled in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Sarit Assouline, MD, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Mazewski C, Platanias LC. A novel approach to overcome drug resistance in acute myeloid leukemia. Haematologica. 2023 Nov 1;108(11):2889-2890. doi: 10.3324/haematol.2023.283099. No abstract available. PMID 37165841
- [Derived] Assouline S, Gasiorek J, Bergeron J, Lambert C, Culjkovic-Kraljacic B, Cocolakis E, Zakaria C, Szlachtycz D, Yee K, Borden KLB. Molecular targeting of the UDP-glucuronosyltransferase enzymes in high-eukaryotic translation initiation factor 4E refractory/relapsed acute myeloid leukemia patients: a randomized phase II trial of vismodegib, ribavirin with or without decitabine. Haematologica. 2023 Nov 1;108(11):2946-2958. doi: 10.3324/haematol.2023.282791. PMID 36951168